CLINICAL TRIAL: NCT07354607
Title: Effect of Transcutaneous Electrical Stimulation on Peripheral Blood Flow - a Pilot Study
Brief Title: Effect of Transcutaneous Electrical Stimulation on Peripheral Blood Flow
Acronym: VASC-STIM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Metropole Savoie (Other)
Collaborators: Laboratoire Interuniversitaire de Biologie de la Motricité (Other); Université Savoie Mont Blanc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHMS25010; 2025-A02335-44 (Other: RCB)
Record Dates: First submitted 2025-12-30; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Volunteer; Adult
Keywords: transcutaneous electrical nerve stimulation; blood flow
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): transcutaneous electrical nerve stimulation
  Interventions: Other: transcutaneous electrical nerve stimulation

INTERVENTIONS:
Other: transcutaneous electrical nerve stimulation — transcutaneous electrical nerve stimulation on arm. 6 different protocol will be apply testing different modality of frequency and positionnement of electrodes

SUMMARY:
The goal of this clinical trial is to learn if transcutaneous electrical nerve stimulation can affect blood flow in healthy volunteers. The main question it aims to answer is:

Determine the stimulation parameters (frequency in the range 5- 100Hz and proximal or distal placement) inducing the most significant hyperaemic response in volunteers.

Participants will attend to one visit ( 1h30) , 6 protocol of stimulation will be tested on his arm . If his agree, an optionnal measure will be made during another visit. During this optionnal visit, two modalities of intensity adjustment will be tested in regard of the result of the first part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged 18 years or older
* Having freely given written consent, after being informed of the purpose of the study, its conduct and its risks.
* Affiliated with a social security scheme

Exclusion Criteria:

* Persons with pacemakers or any other implantable electrical devices,
* Pregnant women
* Suffering from dermatological conditions or muscle/skin lesions on the arms and forearms.
* Participant unable to give free and informed consent.
* Participant unable to comply with the specific procedures of the study.
* Participant deprived of liberty or benefiting from legal protection measures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
stimulation parameters that induce the most significant hyperaemic response | from enrollment to the end of the procedure (1h30)
  Determine the stimulation parameters (frequency in the range 5- 100Hz and proximal or distal placement) that induce the most significant hyperaemic response in volunteers.

SECONDARY OUTCOMES:
Assess the score on a scale of disconfort level during stimulation for each condition | during testing procedure
  The outcome will be assess using a visual analogic disconfort scale ranging from 0 (no disconfort) to 10 (the highest disconfort imaginable).
Compare stimulation intensities between each condition | during testing procedure
Compare muscle metabolic demand between each condition | during testing procedure

OTHER OUTCOMES:
ancillary : Compare blood flow kinetics during long-term stimulation (1 hour) according to the modalities of intensity adjustment over time (no adjustment vs. adjustment). | during testing procedure (second visit)
ancillary : Compare the comfort reported by participants during long-term stimulation based on the methods used to adjust intensity over time (no adjustment vs. adjustment). | during testing procedure (second visit)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Métropole Savoie, Chambéry, France

IPD SHARING:
Plan to Share IPD: Undecided
exploratory research at this time